CLINICAL TRIAL: NCT05035784
Title: Retrograde Colonic Enema With Fecal Microbiota Transplantation vs Retrograde Colonic Enema Only in the Treatment of Childhood Constipation
Brief Title: RCE With FMT in the Treatment of Childhood Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shucheng Zhang, professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A333--1
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Fecal Microbiota Transplantation; Constipation - Functional

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal supernatant (Active Comparator): Fecal supernatant is used for treatment of childhood Constipation
  Interventions: Drug: Fecal supernatant
- non-Fecal supernatant (Placebo Comparator): Placebo is used for treatment of childhood Constipation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fecal supernatant — Fecal supernatant from a child registered in the specimen bank that matches the subject's age, gender, and weight .
  Arms: Fecal supernatant
Drug: Placebo — a placebo designed to match the FMT+RCE group based on appearance including 0.9% physiological saline.
  Arms: non-Fecal supernatant

SUMMARY:
Constipation is the most common complaint in childhood gastrointestinal disease, affecting an estimated 20% of the global children.The treatment strategies consist of diet control, behavioral intervention and oral and sometimes rectal laxatives. Given higher success rate and fewer side effects, the laxative PEG3350 has been considered the first choice in childhood constipation.However, effectiveness of PEG 3350 laxative is not lasting, and the use of PEG increases the risk of fecal incontinence. Additional treatment interventions are still necessary.Enema can act directly on the rectum and distal colon to quickly relieve symptoms of fecal impaction which is considered one of main source of intractable constipation. Children with fecal impaction who received enema had fewer fecal incontinence and diarrhea than children who received PEG. There have been lots of evidence that enema is effective in fecal impaction in children with functional constipation.But there are still cases of recurrences noted after enema. Fecal bacteria transplantation (FMT) is a new treatment method emerging in recent years, which is widely used in the treatment of functional gastrointestinal diseases. FMT has been proved to play a very prominent role in correcting intestinal flora disorders. By transplanting exogenous flora into the intestinal tract of patients, FMT can inhibit bacterial reproduction, regulate intestinal environment and cascade the body immunity, so as to achieve the therapeutic effect of disease.

Retrograde colonic enema with FMT, an new method, provides the possibility for the treatment of childhood constipation. However, there is still a lack of evidence-based support for the treatment of childhood constipation by retrograde colonic enema with FMT. Therefore, we designed a randomized, controlled, double-blind clinical trial to confirm the efficacy and safety of retrograde colonic enema with FMT in the treatment of childhood constipation.

ELIGIBILITY:
Inclusion criteria:

* 4-14 years old;
* Roman IV criteria for childhood constipation;
* After a course of PEG and a course of Chinese medicine treatment was ineffective;
* Barium enema showing fecal impaction.

Exclusion criteria:

* Congenital and/or acquired intestinal diseases, such as congenital megacolon, intestinal stenosis, polyps, Crohn's disease, tuberculosis, inflammation, and tumors;
* Anorectal diseases, such as anal atresia, fistula, abscess, and tumor;
* Neurological diseases, such as brain and spinal cord diseases;
* genetic metabolic diseases;
* psychosocial and behavioral diseases;
* other systemic diseases;
* Refused to participate in.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
improvement of spontaneous bowel movements(SBMs) per week | Baseline
  the frequency of defecation without drugs or other auxiliary methods
improvement of spontaneous bowel movements(SBMs) per week | at the end of 4-weeks FMT treatment
  the frequency of defecation without drugs or other auxiliary methods
improvement of spontaneous bowel movements(SBMs) per week | at the end of 12 weeks follow-up
  the frequency of defecation without drugs or other auxiliary methods
Satisfaction with bowel function | Baseline
  Satisfaction with bowel function was collected from the parents and defined as whether they were satisfied with bowel function after the treatment (yes or no).
Satisfaction with bowel function | at the end of 4-weeks FMT treatment
  Satisfaction with bowel function was collected from the parents and defined as whether they were satisfied with bowel function after the treatment (yes or no).
Satisfaction with bowel function | at the end of 12 weeks follow-up
  Satisfaction with bowel function was collected from the parents and defined as whether they were satisfied with bowel function after the treatment (yes or no).

SECONDARY OUTCOMES:
Bowel movements | Baseline
  the frequency of bowel movements per week
Bowel movements | at the end of 4-weeks FMT treatment
  the frequency of bowel movements per week
Bowel movements | at the end of 12 weeks follow-up
  the frequency of bowel movements per week
Painful or hard bowel movements | Baseline
  The feelings of children during defecation
Painful or hard bowel movements | at the end of 4-weeks FMT treatment
  The feelings of children during defecation
Painful or hard bowel movements | at the end of 12 weeks follow-up
  The feelings of children during defecation
Large diameter or scybalous stools | Baseline
  appearance and wetness of stool
Large diameter or scybalous stools | at the end of 4-weeks FMT treatment
  appearance and wetness of stool
Large diameter or scybalous stools | at the end of 12 weeks follow-up
  appearance and wetness of stool
Excessive volitional stool retention | Baseline
  The number of children who intentionally control or reduce the frequency of defecation
Excessive volitional stool retention | at the end of 4-weeks FMT treatment
  The number of children who intentionally control or reduce the frequency of defecation
Excessive volitional stool retention | at the end of 12 weeks follow-up
  The number of children who intentionally control or reduce the frequency of defecation
Encopresis | Baseline
  the frequency of fecal incontinence
Encopresis | at the end of 4-weeks FMT treatment
  the frequency of fecal incontinence
Encopresis | at the end of 12 weeks follow-up
  the frequency of fecal incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Background] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Background] Gurram B, Sue PK. Fecal microbiota transplantation in children: current concepts. Curr Opin Pediatr. 2019 Oct;31(5):623-629. doi: 10.1097/MOP.0000000000000787. PMID 31169545
- [Background] Xu D, Chen VL, Steiner CA, Berinstein JA, Eswaran S, Waljee AK, Higgins PDR, Owyang C. Efficacy of Fecal Microbiota Transplantation in Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2019 Jul;114(7):1043-1050. doi: 10.14309/ajg.0000000000000198. PMID 30908299
- [Background] Tian H, Ding C, Gong J, Ge X, McFarland LV, Gu L, Wei Y, Chen Q, Zhu W, Li J, Li N. Treatment of Slow Transit Constipation With Fecal Microbiota Transplantation: A Pilot Study. J Clin Gastroenterol. 2016 Nov/Dec;50(10):865-870. doi: 10.1097/MCG.0000000000000472. PMID 26751143
- [Background] Ohkusa T, Koido S, Nishikawa Y, Sato N. Gut Microbiota and Chronic Constipation: A Review and Update. Front Med (Lausanne). 2019 Feb 12;6:19. doi: 10.3389/fmed.2019.00019. eCollection 2019. PMID 30809523
- [Background] Kassam Z, Dubois N, Ramakrishna B, Ling K, Qazi T, Smith M, Kelly CR, Fischer M, Allegretti JR, Budree S, Panchal P, Kelly CP, Osman M. Donor Screening for Fecal Microbiota Transplantation. N Engl J Med. 2019 Nov 21;381(21):2070-2072. doi: 10.1056/NEJMc1913670. Epub 2019 Oct 30. No abstract available. PMID 31665572
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Background] Vriesman MH, Koppen IJN, Camilleri M, Di Lorenzo C, Benninga MA. Management of functional constipation in children and adults. Nat Rev Gastroenterol Hepatol. 2020 Jan;17(1):21-39. doi: 10.1038/s41575-019-0222-y. Epub 2019 Nov 5. PMID 31690829
- [Background] Clemente MG, Mandato C, Poeta M, Vajro P. Pediatric non-alcoholic fatty liver disease: Recent solutions, unresolved issues, and future research directions. World J Gastroenterol. 2016 Sep 28;22(36):8078-93. doi: 10.3748/wjg.v22.i36.8078. PMID 27688650
- [Background] Woodworth MH, Carpentieri C, Sitchenko KL, Kraft CS. Challenges in fecal donor selection and screening for fecal microbiota transplantation: A review. Gut Microbes. 2017 May 4;8(3):225-237. doi: 10.1080/19490976.2017.1286006. Epub 2017 Jan 27. PMID 28129018
- [Background] Vindigni SM, Surawicz CM. Fecal Microbiota Transplantation. Gastroenterol Clin North Am. 2017 Mar;46(1):171-185. doi: 10.1016/j.gtc.2016.09.012. PMID 28164849
- [Background] Shen ZH, Zhu CX, Quan YS, Yang ZY, Wu S, Luo WW, Tan B, Wang XY. Relationship between intestinal microbiota and ulcerative colitis: Mechanisms and clinical application of probiotics and fecal microbiota transplantation. World J Gastroenterol. 2018 Jan 7;24(1):5-14. doi: 10.3748/wjg.v24.i1.5. PMID 29358877
- [Background] Dai M, Liu Y, Chen W, Buch H, Shan Y, Chang L, Bai Y, Shen C, Zhang X, Huo Y, Huang D, Yang Z, Hu Z, He X, Pan J, Hu L, Pan X, Wu X, Deng B, Li Z, Cui B, Zhang F. Rescue fecal microbiota transplantation for antibiotic-associated diarrhea in critically ill patients. Crit Care. 2019 Oct 21;23(1):324. doi: 10.1186/s13054-019-2604-5. PMID 31639033
- [Derived] Gu X, Yang Z, Kou Y, Yang F, Wang Y, Chen Y, Wang E, Jiang X, Bai Y, Zhang Z, Zhang S. Effects of Retrograde Colonic Enema-Based Fecal Microbiota Transplantation in the Treatment of Childhood Constipation: A Randomized, Double-Blind, Controlled Trial. Am J Gastroenterol. 2024 Nov 1;119(11):2288-2297. doi: 10.14309/ajg.0000000000002958. Epub 2024 Jul 11. PMID 38989869